CLINICAL TRIAL: NCT02829099
Title: A Phase 1, Open-Label Study of the Safety, Pharmacokinetics and Pharmacodynamics of JNJ-64457107, an Agonistic Human Monoclonal Antibody Targeting CD40 in Patients With Advanced Stage Solid Tumors
Brief Title: A Study of Safety, Pharmacokinetics and Pharmacodynamics of JNJ-64457107 in Participants With Advanced Stage Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR108186; 64457107CAN1001 (Other: Janssen Research & Development, LLC); 2016-000969-23 (EudraCT Number)
Record Dates: First submitted 2016-07-07; First posted 2016-07-12 (Estimated); Last update posted 2022-10-06 (Actual); Status verified 2022-10

CONDITIONS: Advanced Solid Neoplasms
MeSH Terms: interventions — mitazalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- JNJ-64457107 (Experimental): In Part 1, the first cohort will receive JNJ-64457107 at a starting dose of 75 microgram per kilogram (mcg/kg). The proposed treatment schedule is intravenous (IV) dosing every 14 days. JNJ-64457107 doses will be escalated following a modified Continual Reassessment Method (mCRM); the JNJ-64457107 dose will be increased by not more than half-logarithmical (3.2-fold) dose increments. Dose escalation will continue until the maximum tolerated dose (MTD) and/or RP2D of JNJ-64457107 are defined or the maximum-administered dose (MAD) has been reached. In Part 2, subjects will receive JNJ-64457107 at the RP2D and regimen determined in Part 1.
  Interventions: Drug: JNJ-64457107

INTERVENTIONS:
Drug: JNJ-64457107 — JNJ-64457107 administered by IV infusion on Day 1 and 14 of a 28-day cycle.
  Other Names: ADC1013

SUMMARY:
The primary purpose of the study is to determine the recommended Phase 2 dose (RP2D) and schedule of JNJ-64457107 when administered intravenously (IV) to participants with advanced stage solid tumors in Part 1 and to further characterize the safety of JNJ-64457107 when administered IV to participants with non-small cell lung cancer (NSCLC), pancreatic cancer and cutaneous melanoma in Part 2.

DETAILED DESCRIPTION:
This study has 2 parts: Dose Escalation (part 1) and Dose Expansion (part 2) which are conducted in 3 phases: Screening Phase (up to 28 days prior to first dose of study drug and includes procedures like electrocardiogram [ECG], serum pregnancy test), Treatment phase (continues until the completion of the End-of-Treatment Visit [30 days after last dose of study drug]) and Post-treatment follow-up phase (continues until the participant has died, is lost to follow-up, or has withdrawn consent or the study ends). In follow-up, participants will continue to be monitored for survival status and subsequent cancer-related therapies until the end of study. Additional bio-markers will be assessed, in an optional sub-study, to define the impact of JNJ-64457107 on innate and adaptive immune responses in tumors. Safety will be monitored throughout the study by Safety Evaluation Team (SET).

ELIGIBILITY:
Inclusion Criteria:

* Part 1: advanced stage solid tumors; Part 2: non-small cell lung cancer (NSCLC), pancreatic cancer and cutaneous melanoma
* Eastern cooperative oncology group (ECOG) performance score of 0 or 1
* Adequate organ function as defined in the protocol
* A woman of childbearing potential must have a negative highly sensitive serum (beta-human chorionic gonadotropin [beta-hCG]) pregnancy test at Screening and a negative urine pregnancy test prior to the first dose of study drug
* During the study and for at least 120 days after receiving the last dose of study drug, in addition to the highly effective method of contraception, a man who is sexually active with a woman of childbearing potential must agree to use a barrier method of contraception (example [eg.], condom with spermicidal foam/gel/film/cream/suppository), or who is sexually active with a woman who is pregnant must use a condom

Exclusion Criteria:

* Malignancy other than the disease under study within 2 years before screening (exceptions are squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix, or malignancy that in the opinion of the investigator, with concurrence with the sponsor's medical monitor, is considered cured with minimal risk of recurrence)
* Symptomatic brain metastases; asymptomatic brain metastases are allowed provided that they have been treated, have been stable for greater than (>) 6 weeks as documented by radiographic imaging, and do not require prolonged (>14 days) systemic corticosteroid therapy
* Treatment with any local or systemic anti-neoplastic therapy or investigational anticancer agent within 14 days or 4 half-lives, whichever is longer, up to a maximum wash-out period of 28 days prior to the initiation of study drug administration
* Toxicities from previous anti-cancer therapies have not resolved to baseline levels or to Grade 1 or less except for alopecia and peripheral neuropathy
* Major surgery (eg., requiring general anesthesia) within 3 weeks before screening, or will not have fully recovered from surgery, or has surgery planned during the time the subject is expected to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2016-09-21 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-29 (Actual)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicities (Part 1) | Up to 28 days
  Dose-limiting toxicities will be reviewed as a subset of adverse events that occur within the first 28 days of dosing and meet protocol-specified criteria.
Incidence of adverse events (Part 1 and 2) | From signing of informed consent form (ICF) until 30 days after last dose of study drug (approximately up to 29 Months)

SECONDARY OUTCOMES:
Overall response rate (ORR) | Disease assessment will continue until progression or lost to follow-up (approximately up to 29 months)
  The ORR is the proportion of participants with confirmed best objective response of complete response (CR) or immune-related CR (irCR).
Duration of Response (DOR) | Disease assessment will continue until progression or lost to follow-up (approximately up to 29 months)
  For participants who achieve CR or partial response (PR), DOR will be calculated as time from initial response of CR or PR to progressive disease or death due to underlying disease, whichever comes first.
Progression-free Survival (PFS) | Disease assessment will continue until progression or lost to follow-up (approximately up to 29 months)
  PFS is defined as the time from first dose of JNJ-64457107 to progressive disease or death due to any cause, whichever occurs first.
Overall Survival (OS) | Disease assessment will continue until progression or lost to follow-up (approximately up to 29 months)
  Overall survival is defined as the time from first dose of JNJ-64457107 to date of death from any cause.
Maximum observed serum concentration (Cmax) of JNJ-64457107 | Cycle 1 Day 1 and Cycle 2 Day 15: predose, 1, 4, 24, 48, 72 hours post end of infusion (EOI); any time (Cycle 1 Day 8 and Cycle 2 Day 22); predose (Cycle 1 Day 15 and Cycle 3 and 4); end of treatment
Time of maximum observed serum concentration (Tmax) of JNJ-64457107 | Cycle 1 Day 1 and Cycle 2 Day 15: predose, 1, 4, 24, 48, 72 hours post end of infusion (EOI); any time (Cycle 1 Day 8 and Cycle 2 Day 22); predose (Cycle 1 Day 15 and Cycle 3 and 4); end of treatment
  The Tmax is defined as actual sampling time to reach maximum observed analyte concentration.
Area under the serum concentration versus time curve from time 0 to infinity (AUCinf) of JNJ-64457107 | Cycle 1 Day 1 and Cycle 2 Day 15: predose, 1, 4, 24, 48, 72 hours post end of infusion (EOI); any time (Cycle 1 Day 8 and Cycle 2 Day 22); predose (Cycle 1 Day 15 and Cycle 3 and 4); end of treatment
  The AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time, calculated as the sum of AUC(last) and C(last)/lambda(z); wherein AUC(last) is area under the plasma concentration-time curve from time zero to last quantifiable time, C(last) is the last observed quantifiable concentration, and lambda(z) is elimination rate constant.
Area under the serum concentration versus time curve from time 0 to the final quantifiable time point (t) [AUC(0-t)] of JNJ-64457107 | Cycle 1 Day 1 and Cycle 2 Day 15: predose, 1, 4, 24, 48, 72 hours post end of infusion (EOI); any time (Cycle 1 Day 8 and Cycle 2 Day 22); predose (Cycle 1 Day 15 and Cycle 3 and 4); end of treatment
Area under the serum concentration versus time curve during a dosing interval (AUCtau) of JNJ-64457107 | Cycle 1 Day 1 and Cycle 2 Day 15: predose, 1, 4, 24, 48, 72 hours post end of infusion (EOI); any time (Cycle 1 Day 8 and Cycle 2 Day 22); predose (Cycle 1 Day 15 and Cycle 3 and 4); end of treatment
Immunogenicity of JNJ-64457107 when administered IV | Cycle 1: predose on Day 1; Cycle 2: predose on Day 1; Cycles 3, 4: predose; end of treatment visit
  Detection and characterization of antibodies to JNJ-64457107

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (4):
- Israel (3):
  - Haifa
  - Jerusalem
  - Tel Aviv
- Madrid, Spain

REFERENCES:
- [Derived] Andersson H, Sobti A, Jimenez DG, de Coana YP, Ambarkhane SV, Hagerbrand K, Smith KE, Lindstedt M, Ellmark P. Early Pharmacodynamic Changes Measured Using RNA Sequencing of Peripheral Blood from Patients in a Phase I Study with Mitazalimab, a Potent CD40 Agonistic Monoclonal Antibody. Cells. 2023 Sep 27;12(19):2365. doi: 10.3390/cells12192365. PMID 37830579
- [Derived] Moreno V, Perets R, Peretz-Yablonski T, Fourneau N, Girgis S, Guo Y, Hellemans P, Verona R, Pendas N, Xia Q, Geva R, Calvo E. A phase 1 study of intravenous mitazalimab, a CD40 agonistic monoclonal antibody, in patients with advanced solid tumors. Invest New Drugs. 2023 Feb;41(1):93-104. doi: 10.1007/s10637-022-01319-2. Epub 2022 Dec 20. PMID 36538259